CLINICAL TRIAL: NCT02481076
Title: Compression in Anklefracture Treatment, The CAT-study
Acronym: CAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hillerod Hospital, Denmark (Other)
Collaborators: The Research Unit, Northzealand Hospital (Unknown); Department of Orthopedic Surgery, Northzealand Hospital (Unknown)
Responsible Party: Principal Investigator, Rikke Winge, PhD-student, MD, Hillerod Hospital, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-2-2013-140
Record Dates: First submitted 2013-10-08; First posted 2015-06-25 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Ankle Fractures
Keywords: malleolar fractures; ORIF; compression; infection; wound dehisence
MeSH Terms: conditions — Ankle Fractures; Infections | interventions — Compression Bandages

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- compression therapy (Experimental): Intervention arm: administration of
  * Flowtron Hydroven boot in the Emergency Department
  * Coban2 Lite after surgery
  * Flowtron Hydroven boot after surger, before discharge
  Interventions: Device: Flowtron Hydroven and Coban2 Lite; Device: compression bandage
- controle (Other): The leg is elevated on a Braun frame. This is the "old fashioned" conservative treatment to prevent swelling.
  Interventions: Other: Braun frame

INTERVENTIONS:
Device: Flowtron Hydroven and Coban2 Lite — The patient in the intervention group will use both compression boot and compression bandage, as described in intervention arm
  Other Names: Flowtron Hydroven; Coban2 Lite
  Arms: compression therapy
Other: Braun frame — The leg is elevated on a Braun frame
  Arms: controle
Device: compression bandage — application of flowtron hydroven boot and compression bandage
  Arms: compression therapy

SUMMARY:
The aim of this project is to find out if compression treatment can lower the incidens of surgical wound complications, such as infection and wound rupture, in patients with ankle fractures. The compression regime consists of a two-layered compression stocking applied after surgery and a massage boot applied both before and after surgery.

The largest part of the study is the clinical trial, with which we aim to prove the hypothesis:

* That the compression regime reduces wound infections from 10-40% to 5% on patients with a broken ankle (Either one side of the ankle, two or three sides (including the posterior part of the ankle))

DETAILED DESCRIPTION:
Malleolar fractures

Surgical treatment of patients with malleolar fractures imposes a special challenge for orthopaedic surgeons. A typical ankle fracture results in haematoma, sometimes blistering and almost always oedema formation. This postpones the optimal time for surgery. When operating on a swollen ankle, it becomes obvious for the surgeon that the tissue elasticity and normal structure is changed. This can complicate the surgical approach, procedure, the reduction of the fracture and the closure of the incision. Quite often the skin is difficult to adapt, resulting in excessive tension on the sutures. This can potentially lead to skin necrosis and wound dehiscence. Blood and fluid imbibed tissue and prolonged operating time, increases the risk of post-operative infection, and thereby give the patient painful and extended post-operative course.

When striving to give the patient a good treatment and rehabilitation, it is paramount to prevent surgical complications.

Compression therapy, as part of the standard treatment of ankle fractures, is not yet described in the literature and no previous study has tested its efficiency in this patient group, in a systematic manner. It is a new, innovative way of helping the patients to faster rehabilitation and to prevent surgical soft tissue complications.

If this study proves the expected effect on soft tissue complications, compression therapy will probably also show an effect on other fracture types: knee-, wrist-, tibia- and femoral fractures, making compression therapy an integrated part of the standard fracture regime in all orthopaedic departments.

Malleolar fractures in Denmark has an incidence of 107/100.000 person, making it one of the most common fracture types in the country. In Denmark 6000 malleolar fractures are operated each year.

Studies have shown increased complication rates in the elderly, diabetics, smokers, patients on immunomodulating medication, alcoholics, and patients with osteoporosis and peripheral neuropathy.

Treatment of malleolar fractures in Denmark shows great local variations, and standard differs between hospitals, often with a low grade of clinical evidence.

Nordsjællands Hospital has decided, to implement a standard regime of Flowtron Hydroven 3™ and Coban™ 2 lite, to prevent oedema formation and blistering. The decision came after clinicians having observed a high incidence of oedema, blistering and wound healing problems in this cohort of patients, often forcing surgeons to postpone surgery and prolonging inpatient stay, resulting in a long and cumbersome rehabilitation for the patient.

Intermittent pneumatic compression

Intermittent pneumatic compression (IPC) is used mainly in prevention of DVT. The use of IPC in treatment of postoperative soft tissue care is only sporadically mentioned in the literature. These studies define the mechanisms of action as either mechanical or chemical. The mechanical effect is due to improved vascularity, redirection of blood flow and cyclic loading. The chemical effect is caused by increased production of nitric oxide (NO), producing vasodilation and the increase of inflammatory mediators, promoting heeling by stimulating proliferation of fibroblasts and endothelial cells. Some studies have investigated the effect of IPC on the vascularity of bone and soft tissue (animal studies), fracture related oedema and oedema related to venous disease and other medical conditions, showing a convincing effect on all. Accumulating data from experimental animal studies suggest that the use of IPC increases neurovascular ingrowth, the amount of newly organized parallel collagen fibres, fibroblast proliferation and proliferative repair. Further IPC counteract the negative influence immobilization has on tissue repair. Therefore, theoretically one should expect that application of an IPC unit on a newly operated and immobilized patients ankle, would prevent oedema formation, speed up tissue regeneration and enhance arterial blood flow thereby preventing wound healing problems defined as infection, wound dehiscence, prolonged healing, skin necrosis, exposed hardware, and maybe also accelerate bone heeling.

COBAN 2 lite

Coban™ 2 lite is a compression bandage consisting of an inner comfort layer and an outer stretch layer, designed to deliver therapeutic compression for the treatment of venous leg ulcers and related conditions. The bandage is purposed for patients less tolerant of compression, with mixed aetiology and a ABPI (ankle brachial pressure index) ≥ 0,5. Correctly applied, the bandage take the form of a solid tube which reduces slippage and let the patient wear it for up to several weeks without the need of re-application. The use of compression stockings and bandages are well described in literature, and an integrated part of the management of oedema end venous ulcers, but not addressed when it comes to fracture treatment.

Adverse effects

Intermittent pneumatic compression The IPC device is routinely employed in prevention of deep venous thromboembolism (DVT) and subsequently pulmonary embolism (PE) and in the management of lymfoedema. It is considered a safe and efficient alternative to medical thromboprophylaxis and only few adverse effects have been described in literature, all consisting of case reports.

When using IPC as DVT prophylaxis it is often applied during surgery and with the patient in general anaesthesia, hindering the patient in reporting any discomfort. One author describes a case, where application of IPC on a patient with cancer associated thrombosis and embolism, results in a pulmonary embolism. The patient did not show signs of having a DVT prior to surgery, and the author concludes that the PE might have taken place regardless of the application of IPC devices.

Two case reports describes peroneal nerve palsy as a possible adverse effect to IPC. The first case concerns a woman with pancreatic cancer and weight loss, who develops peroneal nerve palsy bilaterally under surgery, probably because there is no subcutaneous fat to protect the nerve against the applied pressure between the fibular head and the compression boot. The second case concerns an obese patient undergoing 10 hours intracranial surgery.

One author reports a case where an older woman with postoperative delirium and fragile skin develops hemorrhagic bullae under the IPC-device. This could probably have been avoided, had the patient not ben delirious an inept of reporting discomfort.

Some authors have tried to associate the IPS unit to compartment syndrome, but the cases have all been on patients whom have undergone prolonged operation in the lithotomy state, which is known to increase the risk for compartment syndrome in the lower leg.

Malfunctioning of the equipment is described in literature, but is rare. The IPC-device can cause warmth and sweating under the inflatable textile and discomfort if it is placed incorrectly or directly on top of a suture.

Compression bandage

There are no descriptions in literature of major side effects to the compression bandage. During the early implementation of compression treatment of malleolar fracture at the unit of Orthopaedic Surgery, Nordsjællands Hospital, pressure-wounds have been observed, and in one case with a visible Achilles tendon. Several minor pressure wounds have been noted, but these have all successfully healed under conservative treatment.

The Coban™ 2 lite can cause discomfort such as tightness, if applied to firmly. The inner comfortlayer can chafe bony prominences or tendons if applied to thick.

Precautionary measures

In order to prevent any side effects or discomfort, the project manager routinely and frequently examines all patients included in the trial. This will take place both in the Emergency Department, at the bedward 48-72 hours after admission, and postoperatively.

The staff will receive ongoing training in the application and observation of both Coban™ 2 lite and the Flowtron Hydroven 3™, in order to prevent any malfunctioning or misapplication.

Hypotheses and Aims

Hypotheses

Study1 - That the compression regime reduces wound infections from 10-40% to 5% on patients with mono-, bi-, and trimalleolar fractures treated according to the ORIF-principles (open reduction internal fixation)

Study 2

- That the retrospective study will establish the historical incidence of infections, before the compression regime was implemented.

Study 3 - That a systematic literature review will reveal the extent of infection and provide the author with knowledge of regimes described in international literature, aiming at lowering the incidence of infections.

Aims

Study 1

* To perform a prospective, un-blinded, controlled cohort study, to evaluate the effect of Flowtron Hydroven3™ and Coban2 lite™ on the incidence of complications (infection, wound dehiscence, prolonged healing, skin necrosis, exposed hardware, DVT, amputation and death) after operation for mono-, bi- and trimalleolar fractures at Nordsjællands Hospital.
* Study 2

To perform a retrospective evaluation of the treatment for mono-, bi- and trimalleolar fractures, at Nordsjællands Hospital, Department of Orthopaedic Surgery, before the current compression management was implemented, focusing on the following parameters:

A) Pre-operative compression/deflating management (elevation, Flowtron Hydroven™), prevalence of oedema, blistering, smoking, diabetes, co-morbidity, age and sex)

B) Per-operative parameter: administration of antibiotics.

C) Postoperative compression/deflation management (elevation, Flowtron Hydroven™ og Coban2 lite™ ), oedema, blistering, infection, wound dehiscence, prolonged healing, skin necrosis, exposed hardware, DVT, amputation and death.

- Study 3 To perform a literature study, enabling the author to describe, and establish the incidence of surgical complications for mono-, bi- and trimalleolar fractures, resulting in a review article.

Project Plan

The study is divided into 3 phases:

Sub study 1: A prospective, mono-centre, randomized, controlled, non-blinded, cohort study, with a postoperatively follow-up period of 6 weeks.

Sub study 2: A retrospective, mono-centre, cohort study based on patient files, with follow-up period of 6 weeks from the day of operation.

Sub study 3: A literature study.

Study period

Sub study 1: 1.11.2013 - 5.12.2015 Sub study 2: 1.10.2013 - 1.5.2015 Sub study 3: 1.10.2013 - 1.10.2014

Study population

* Sub study 1: Each year approximately 170 patients are operated on for mono-, bi- and trimalleolar fractures. According to the power calculation (2x78)= 156 patients needs to be included in the study group. The inclusion period will run for 24 months, or till 156 patients are included.
* Sub study 2: All patients operated for mono-, bi- and trimalleolar fractures, in a 12 months period (1/1/2009-31/12/2009) before implementing the compression treatment consisting of Flowtron Hydroven™ and Coban2 lite™ the unit of Orthopaedic surgery, Nordsjællands Hospital.
* Sub study 3: Literature search on PubMed, on patients with ankle fractures, operated according to ORIF. Search words: ankle fracture/malleolar fracture, ORIF, complications, infections, wound dehiscence, necrosis and amputation.

Language: English.

Data sources:

InfoView:

A datawarehouse database containing CPR-numbers coupled to SKS-codes (Sundhedsvæsenets Klassifikations System, diagnosis codes). All patient contact to the Emergency Department, Out Patient Clinic and bed wards are recorded here.

OPUS:

IT-system containing the patient files necessary to perform sub study 2.

Centricity:

IT-system containing x-rays. Will be used to identify and classify ankle fractures on the patients whose data are found via InfoView.

Labka:

A system contained in OPUS, where blood sample-results are kept.

Orbit:

IT-system doctors use to book patients for surgical procedures, used to find all surgical procedures for a given code, a given year.

PubMed:

Database accessing primarily the Medline database of references and abstracts on life sciences and biomedical topics.

Procordo

Randomization, stratification, visualization of data, and data storage will be managed using an IT system called Procordo (Procordo ApS Rugaardsvej 5 DK-8680 Ry Denmark).

Study procedures

Study design:

Sub study 1: Patients are included in the Emergency Department (red) by the doctor on duty or the project manager, if they are willing to participate and have given consent after written and oral information about the study. As part of the standard treatment, X-rays are taken to confirm the diagnosis. The fracture will be evaluated for the need of surgery, according to the department standard:

1. Unstable fractures (SU3+4, SA2, PA2+3, PU2+3+4). Particularly SU-fractures are important to examine closely, in order to rule out ligamentous damage on the medial malleolar.
2. Dislocated fractures in the lateral malleolus, with maximum diastases of 2 mm.
3. Fracture of the medial malleolus.

Standard blood tests will be carried out, if deemed necessary, and the affected ankle will be treated with a splint, according to the Emergency Department's standard procedures. The patient will hereafter get randomized. Randomization, stratification, visualization of data, and data storage will be managed using an IT system called Procordo (Procordo ApS Rugaardsvej 5 DK-8680 Ry Denmark). Patients will be block randomized into blocks of 6-10. This size is chosen because of the stratification according to two variables, to make sure that an equal distribution of stratae is obtained each block. Block size is blinded for the researcher. The system will use a sequence of 300, and patients will be stratified according to diabetes, smoking and need for closed reduction. The patient will be on-line randomized in the emergency department, as close to the actual treatment as possible, in order to prevent superfluous drop-out. Randomization is handled by either a doctor or a nurse using a computer interface designed by Procordo. The person to include will open the computer, use the shortcut symbol to the randomization interface, type the user name and code accessible to the personnel in the emergency department. A sign with username and code will be hanging next to the computer. The user will be asked to identify him/herself by name, and to type several patient specific parameters: sex, CPR-number, fracture type, diabetes, smoking and others. The computer will search in the 300-sequence and come up with the next available number (either 1 or 2) to allocate the patient. The sequence is designed according to block-size, p-value (0,5 or 0,5) and the total number of 300. The allocation process itself is hidden from the investigator, and at no point in the process, will the system reveal if the patient is in the treatment- or the control-arm. This makes it possible to blind the treatment later on, when the patient visit the out-patient clinic. In theory the randomization interface is accessible to all personnel in the emergency department, which is why every inclusion will be checked by the project manager.

To avert confounding treatments, a sign will be put on the patient bed during hospitalization, communicating which group the patient belongs to.

The project manager will control that the intervention/non-intervention is applied according to the study protocol. This is done by continuous visits to the bed ward, examining the patients to see if the Coban2 lite™, Flowtron Hydroven™ and Braun frame are correctly used.

The Intervention group (pink): Will receive compression therapy in the form of a Flowtron Hydroven™, 40-60 mmHg, ¾-1 hour, 3 times a day, when diagnosed and allocated in the emergency department, either on top of the splint, or if no splint is administered, on top of the dressing. This treatment will be continued, until the patient is fit for surgery according to clinical priority and theatre availability. The surgical procedure will follow the standards of the Department of Orthopaedic Surgery.

After finished surgery, the doctor or nurse in the operating room (OR) will apply a dry, non-adherent, wound dressing (Vliwasorb® Lohmann & Rauscher, Gøngehusvej 252, DK-2950 Vedbæk, Denmark) and Coban2 lite™. The patient will continue the Flowtron Hydroven™ treatment in the bed ward (40-60 mmHg, ¾-1 hour 3 times a day) on top of the Coban2 lite™ bandage, until discharge.

Before discharge the patient is fitted with a Walker boot, unless there is bad compliance or no pulse in arteria dorsalis pedis or tibialis anterior, in which case a CobraCast walking bandage is applied. Both boot and bandage is applied at the bed ward, when the patient has recovered from anaesthesia/analgesia, and worn during fysiotherapy and mobilization. Observation and control of both Flowtron Hydroven™ and Coban2 lite™ in the ward are carried out by the nurses with special training, according to standard procedures, and by the project manager who will collect data between 48-72 hours after admission. On the day of discharge, the Coban2 lite™ is removed, the wound dressing changed and a new Coban2 lite™ is re-applied. According to standard treatment, x-rays are taken after 2 and 6 weeks, and the patient is seen in the outpatient clinic accordingly. At both visits, clinical photos will be taken of the surgical wound, in order to blind the clinical evaluation. Two senior doctors will later be asked to evaluate the photos and determine if infection or wound dehiscence is present. At the 2 weeks visit the Coban2 lite™ and stitches are removed, and a compression stocking is fitted. The project manager will note any wound healing problems (infection, wound dehiscence, skin necrosis, visible osteosynthesis material).

The Walker boot or CobraCast walking splint is re-applied. At the 6 weeks visit, x-rays will be taken, and again the project manager will note any wound healing problems (infection, wound dehiscence, skin necrosis, visible osteosynthesis material). If all parameters are acceptable, the patient course, and follow up is concluded.

The control group: In the Emergency Department the affected leg will be elevated on a Braun Frame, and this treatment will continue in the bed ward, until the patient is fit for surgery according to clinical priority and theatre availability.

The surgical procedure will follow the standards of the Department of Orthopaedic Surgery.

After surgery, a Vliwasorb® wound dressing and TubiGrip™ bandage (Mölnlycke Health Care ApS, Gydevang 33, DK-3450 Allerød, Denmark) is applied. Finally the ankle is stabilized in a Walker boot, unless there is bad compliance or no pulse in arteria dorsalis pedis or tibialis anterior, in which case a CobraCast walking bandage is applied. Both boot and bandage is applied at the bed ward, when the patient has recovered from anaesthesia/analgesia, and worn during fysiotherapy and mobilization. According to standard treatment, x-rays are taken after 2 and 6 weeks, and the patient is seen in the outpatient clinic accordingly. At both visits, clinical photos will be taken of the surgical wound, in order to blind the clinical evaluation. Two senior doctors will be asked to evaluate the photos and determine if infection or wound dehiscence is present. At the 2 weeks visit, the TubiGrip™ and stitches are removed. The project manager will note any wound healing problems (infection, wound dehiscence, skin necrosis, visible osteosynthesis material), and the TubiGrip™ and Walker boot are re-applied. At the 6 weeks visit, X-rays will be taken, and again the project manager will note any wound healing problems (infection, wound dehiscence, skin necrosis, visible osteosynthesis material). If all parameters are acceptable, the patient course, and follow up is concluded.

Sub study 2: All treatments in this study have been closed, at the time of data collection. So the project will have no influence on the course of the patients.

Material:

Sub study 1: Each year approximately 170 malleolar fractures are operated on at Nordsjællands Hospital. Of these 78 are realistically to be included into the project, and studied according to the study variables outlined below. The inclusion period runs for 24 months or till (2x78) = 156 patients are included, and start 1/10/2013.

Sub study 2: The 1/10/2013 the retrospective cohort study begins. 78 patient files will be studied according to the study variables outlined below. The patient files must be dated from before the department of orthopaedic surgery implemented the use of compression therapy as a routine treatment for ankle fractures.

5 Study variables Applies to both, the intervention and control group.

Pre-operative data

* CPR-number
* Age
* Sex
* Smoking at the time of admission (yes/no) (stratification variable)
* Diabetes (yes/no) (stratification variable)
* Alcohol consumption (<1 unit/week, 2-7/14 units/week, >7/14 units/week)
* Need for closed reduction (yes/no) (stratification variable)
* Palpable pulse in foot
* Application of Flowtron Hydroven3 (yes/no) (only intervention group)
* Elevation of on Braun Frame (yes/no) (only control group)
* Fracture date

Per-operative data

* Administration of antibiotics (yes/no)
* Duration of surgery (in minutes)
* Skin blisters of effected leg (pale, red or black. The presence of only one blister from the knee and down results in a positive answer)
* Application of Coban2 Lite after surgery (yes/no) (only intervention group)
* Surgeon's level of training (reservelæge/1. reservelæge/afdelingslæge/overlæge)
* Time from admission (Emergency Department) to surgery (in hours)
* Fracture type (Lauge Hansen)

Post-operative data during hospitalization, collected 48-72 hours after surgery

* Application of Flowtron Hydroven3 (yes/no) (only intervention group)
* Elevation of on Braun Frame (yes/no) (only control group)
* Death (yes/no)
* Adverse effects (pressure soars (type I-IV), peroneal nerve palsy, DVT, pulmonary embolism
* Administration of anticoagulants
* Support on operated leg (yes/no)

Post-operative data collected at the 1st visit to the outpatient clinic, 2 weeks after surgery.

* Date for visit
* Infection (fever, swelling, pain, redness, secretion, need for antibiotics)
* Wound dehiscence (partial or complete rupture of the layers in the wound).
* Skin necrosis (wound edges with pale, black or otherwise non-vital skin)
* Visible osteosynthesis material (no/minor/major)
* Day of discharge (hours after surgery)
* Deep venous thrombosis (confirmed by ultrasound)
* Time from surgery to discharge
* Surgery date
* X-ray acceptable (yes/no)
* Re-admission (yes/no) Cause
* Clinical photos are taken of the surgical wound

Post-operative data collected at the 2nd visit to the outpatient clinic, 6 weeks after surgery.

* Date for visit
* Infection (fever, swelling, pain, redness, secretion, need for antibiotics)
* Wound dehiscence (partial or complete rupture of the layers in the wound).
* Skin necrosis (wound edges with pale, black or otherwise non-vital skin)
* Visible osteosynthesis material (no/minor/major)
* X-ray acceptable (yes/no)
* Surgery date
* Re-admission (yes/no) Cause
* Deep venous thrombosis (confirmed by ultrasound)
* Amputation (yes/no)
* Death (yes/no)
* Clinical photos are taken of the surgical wound

Primary outcome: Infection.

Secondary outcomes: Wound dehiscence, skin necrosis, visible osteosynthesis material, blisters, DVT, amputation, death.

Screening-log:

During the study a screening-log will be kept. All patients who are potential candidates to randomization will be entered into the log.

Ethical considerations

The National Committee on Health Research Ethics:

An application has been forwarded to the Regional Committee on Health Research Ethics, dated 7/12/2012. Application number: 36522

The Danish Data Protection Agency: journal no. 2012-41-1331. Exempted from reporting on the 5th December 2012, as private medical research projects, which must be reported to the National Committee on Health Research Ethics, are no longer required to report to the Danish Data Protection Agency. The project manager is registered as private responsible for the data (Danish: privat dataansvarlig) and undertakes to ensure that the applicable personal data laws for medical research projects are followed by the research group.

Danish Health and Medicines Authority, Pharmacovigilance and Medical Devices Case no. 2012113737. The study is assessed not to require notification according to the regulations for medical equipment § 9, part 1 and therefore does not require reporting to the National Board of Health or the Danish Health and Medicines Authority, Pharmacovigilance and Medical Devices.

Informed consent:

A decision to participate in the research project will be obtained from all patients participating in the study. The decision is made upon due information on the nature, significance, implications and risks of the project and upon receipt of suitable written documentation. It is made voluntarily by a person who is capable of giving his or her consent. The consent shall be in writing, dated and signed, and is obtained in the Emergency Department (ED) The patient will be recruited in the ED as soon as the inclusion diagnosis is made. The initial contact and inclusion will be handled by the doctor on duty or the project manager. He or she will provide the above-mentioned written and oral information. The patients in the ED are examined in small booths, separated by curtains. This provides the necessary privacy to perform a physical examination, but preventing other patients from overhearing conversation can be difficult. Therefor the patient should be offered the possibility to continue the conversation in a quiet interview room. The patient is offered to have an assessor participate in the conversation. All patients must be offered due reconsideration time before making up their minds, this means enough time to talk to the assessor or make a phone call. For practical reasons though, it will be difficult to offer more than 60 minutes reconsideration time, due to the urgent nature of the trauma and the urgent need for surgery. Furthermore the Flowtron Hydroven™ need to be applied relatively quickly after the patient has been diagnosed with the ankle fracture, in order to obtain the best effect. The nature of the intervention is considered non-invasive and with few adverse effect, justifying the relatively short reconsideration time. The Informed consent form must be signed before the patient leaves the ED and the patient can at any time decide to withdraw from the project, without consequence to further treatment.

Good Clinical Practice The local GCP-committee (GCP region Hovedstaden) has been contacted and report that the study is exempted from reporting to the GCP.

Confidentiality:

All personnel involved in the project are bound by professional confidentiality regarding all private data.

The Danish law on "behandling af personoplysninger" (LOV nr. 429 af 31/05/2000) will be adhered to.

Statistics Data will be analysed in collaboration with statistician Tobias Wirenfeldt Klausen. Data will be collected and partially analysed using SPSS (Statistical Product and Service Solutions, 21, IBM)

Based on literature, which shows a complication rate between 10% and 40%, P1 (representing the expected complication rate in the control group), is set to 20% and P2 representing the expected complication rate in the intervention group) to 5%. Using Lehr's formula for calculating a power of 80% and a two-sided significance level at 0,05. The required sample size in each group = 16/(Standard difference)2

Standard difference= 0,454

(calcualtion details to obtain "standard difference" are difficult to show, due to formatting)

Using the Quick formula:

If the power is 80%, the required sample size in each group is:

16/Standard difference= 16/0,454= 77,6 = 78 patients in each group.

Material and Methods

The (IPC)-unit used in this study is a Flowtron Hydroven 3™ (ArjoHuntleigh A/S Vassingerødvej 52 DK-3540 Lynge). It consists of an inflatable textile-boot connected to a pump providing an intermittent pressure between 30-60mmHg.

The compression bandage used in this study is Coban2 lite™ (3M a/s Hannemans Allé 53, 2300 KBH S, Denmark). It consists of an inner comfort layer and an outer stretch layer, designed to give a resting pressure of more than 40mmHg. On standing it will produce a pressure of more than 60mmHg which is the level accepted as the pressure required to counteract venous hydrostatic pressure in the lower leg.

ELIGIBILITY:
Inclusion Criteria:

* All patients operated on Nordsjællands Hospital, department of Orthopaedic surgery, during the inclusion period, for mono-, bi- and trimalleolar fracture, according to the AO-principles.
* Age above 18 years.

Exclusion Criteria:

Sub study 1:

* Age under 18
* Dementia
* Need for external fixation
* Known or suspected DVT or pulmonary embolism
* Patients without Danish CPR-number, or address in Denmark
* Patients who doesn´t want to participate or who are not able to give written or oral consent
* No palpable pulse in the foot in the affected leg (the posterior tibial,- or dorsal artery)
* Multi-traumatized patients and patients with fractures of more than one extremity

Sub study 2:

* Age under 18
* Dementia
* Need for external fixation
* Multi-traumatized patients and patients with fractures of more than one extremity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2013-11; Primary Completion 2015-12 (Actual); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
number of participants with post-surgical wound infection, after ankle fracture operation, | Within the first 6 weeks after surgery.
  The project manager will evaluate the patient twice during the 6 weeks follow-up, in the out-patient clinic. Clinical pictures will be taken at each visit, for two senior doctors to perform a blinded evaluation according to the primary outcome. Infection is defined as Increased pain, swelling, pus secretion, redness, or warmth around the affected area. Need for antibiotics. Not all signs has to be present. The outcome is registred as "number of patients with infection"

SECONDARY OUTCOMES:
Wound dehiscence. | Within the first 6 weeks after surgery.
  Dehisence of the epidermis or the entire dermis. Can be answered with yes/no
Skin necrosis. | Within the first 6 weeks after surgery.
  Pale, dark or non-vital skin, sorrounding the wound.
Visible osteosynthesis material | Within the first 6 weeks after surgery.
  Is the osteosynthesis material visible when the wound is examined or probed during the 2nd. and 6th. week examination in the out-patient clinic. Can be answered with no/yes/a little/ a lot
Blisters | Within the first 6 weeks after surgery.
  Blisters (pale or dark) from the knee and down. Can be answered with yes/no
Deep venous thrombosis | Within the first 6 weeks after surgery.
  Pain, swelling and tenderness in one of the legs, heavy ache in the affected area.
  Warm skin in the area of the clot. Redness of the skin. Elevated D-dimer, confirmation of diagnosis by ultrasound. Can be answered with yes/no
Amputation | Within the first 6 weeks after surgery.
  Amputation og the ankle. Can be answered with yes/no
Death | Within the first 6 weeks after surgery.
  Can be answered with yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Stig Sonne-Holm, Ass. Prof., Study Director — Hvidovre University Hospital
Locations (1):
- Unit of Orthopedic Surgery, Nordsjællands Hospital, Hillerød, Hillerød, Denmark

IPD SHARING:
Plan to Share IPD: No